CLINICAL TRIAL: NCT05656339
Title: Metabolic Effects of Whey Protein Supplementation After Fasting in Volunteers: A Controlled Randomized Crossover Trial
Brief Title: Metabolic Effects of Whey Protein Supplementation After Fasting in Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Mato Grosso (Other)
Collaborators: Univag Centro Universitário (Other)
Responsible Party: Principal Investigator, José Eduardo de Aguilar-Nascimento, MD, PhD, Professor, Federal University of Mato Grosso
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 42481121.3.0000.5692
Record Dates: First submitted 2022-11-22; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Ketosis; Acute-Phase Response; Insulin Resistance
Keywords: Ketone bodies; Whey protein; Fasting
MeSH Terms: conditions — Ketosis; Acute-Phase Reaction; Insulin Resistance; Fasting

STUDY DESIGN:
Intervention Model Description: Male volunteers, aged between 18 and 27 years, healthy, with no report of acute illness during 3 months prior to the study will be included. Individuals with obesity (calculated body mass index above 30 kg/m2), those who reported consumption of alcoholic beverages or any nutritional supplement during the study period will be excluded. The 30 selected volunteers will be scheduled to came to the laboratory after an overnight fast of 12 hours. Participants in the fasting group will immediately collect blood samples. The CHO and the CHO+WP groups will drink 200 ml of the respective supplements described above. After an interval of three hours after ingestion of the supplement, blood samples will be collected again for biochemical assays.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor will not know the randomization nor the phases of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 12 hours Fast - Fast Group (Sham Comparator): Participants will proceed in 12 hours fast condition for blood collection for laboratory assays
  Interventions: Dietary Supplement: Fast
- Carbohydrate plus whey protein supplement - CHO+WP group (Active Comparator): After 12 hours fast participants will collect blood samples and immediately will drink an oral supplement containing carbohydrates plus whey protein. After 3 hours of ingesting the supplement blood samples will be collected again
  Interventions: Dietary Supplement: CHO+WP
- Carbohydrate supplement - CHO group (Placebo Comparator): After 12 hours fast participants will collect blood samples and immediately will drink an oral supplement containing carbohydrates alone without whey protein. After 3 hours of ingesting the supplement blood samples will be collected again
  Interventions: Dietary Supplement: CHO

INTERVENTIONS:
Dietary Supplement: CHO+WP — Oral supplement containing carbohydrates plus whey protein
  Arms: Carbohydrate plus whey protein supplement - CHO+WP group
Dietary Supplement: CHO — Oral supplement containing carbohydrates
  Arms: Carbohydrate supplement - CHO group
Dietary Supplement: Fast — Fast condition of 12 hours
  Arms: 12 hours Fast - Fast Group

SUMMARY:
This study aims to investigate the early metabolic effects and acute phase response of an oral clear supplement containing whey protein plus carbohydrates in young healthy volunteers during fasting-induced organic response

DETAILED DESCRIPTION:
The investigators will enroll young male healthy volunteers. In this controlled crossover clinical trial, after a 12-hour fast, subjects will be randomized to consumed either: a) 200ml of carbohydrates enriched with whey protein (CHO+WP; n=30); or b) 200ml of water plus maltodextrin (CHO group, n=30); or c) remained fasting (Fast group; n=30). Blood samples will be collected after 12h-fast and three hours after the ingestion of the supplements (or 3h fast in Fast group) for blood glucose; glycated hemoglobin; serum insulin; C-reactive protein; beta-hydroxybutyrate; triglycerides; albumin; chlorine and sodium assays. After a temporal break of seven days an inversion of the groups will performed so all subjects entered in the three groups. Group CHO+P will drink a clear non-residual supplement (698 mOsm/L) having 100% whey protein isolated from total proteins, with various vitamins (B1, B6, C, D, niacin and folic acid) with a "lemon tea" flavor (Nutren Fresh; Nestlé, São Paulo, Brazil). The formula contains no lactose or lipids; is formulated with a volume of 200ml, with a caloric density of 1.28kcal/ml; protein: 10g in 200ml of the product (100% whey protein isolate); and carbohydrate: 54g in 200ml of the product (74% glucose syrup and 26% maltodextrin); Group CHO will received a clear supplement containing 200 mL of water combined with unflavored 25 g of 100% maltodextrin (CarboCH - Prodiet, Curitiba, Brazil) at 12.5% dilution (101 mOsm/kg; 95kcal/200ml). The third group (Fast group; n=10) will not consume any food or supplement.

ELIGIBILITY:
Inclusion Criteria:

* Male young healthy volunteers

Exclusion Criteria: or will be excluded.

* Individuals with obesity (calculated body mass index above 30 kg/m2)
* Participants reporting consumption of alcoholic beverages
* Consumption of any nutritional supplement during the study period

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in serum hydroxy butyrate | Change from 12 hours fasting (baseline) at 3 hours after the ingestion of the oral supplement
  Serum hydroxy butyrate levels from 12 hours fast at 3 hours after ingestion of oral supplement
Change in acute phase response proteins | Change from12 hours fasting (baseline) at 3 hours after the ingestion of the oral supplement
  Change of serum C reactive protein and albumin from 12 hours fast (baseline) to 3 hours after ingestion of the oral supplement
Change in insulin resistance | Change from12 hours fasting (baseline) at 3 hours after the ingestion of the oral supplement
  Change of HOMA index from 12 hours fast (baseline) to 3 hours after ingestion of the oral supplement

CONTACTS AND LOCATIONS:
Overall Officials: Jose E Nascimento, MD, PhD, Principal Investigator — Univag Centro Universitário
Locations (1):
- Centro Universitário de Varzea Grande (UNIVAG), Várzea Grande, Mato Grosso, Brazil

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with researchers that contact with the investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year
Access Criteria: email do jose.aguilar@univag.edu.br